CLINICAL TRIAL: NCT06731452
Title: Exploring Markers of Brain Health With EEG and TMS: A Pilot Study
Brief Title: Exploring Neurophysiological Markers of Brain Health
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas at Dallas (Other)
Responsible Party: Principal Investigator, Sandra Chapman, PhD, Professor, Chief Director of UTD Center for BrainHealth, The University of Texas at Dallas
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 24-315
Record Dates: First submitted 2024-12-05; First posted 2024-12-12 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Healthy Lifestyle; Health-Related Behavior
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Online Strategic Memory Advanced Reasoning Training & Stress Solutions (Experimental): Strategic Memory Advanced Reasoning Training (SMART) teaches meta-cognitive strategies for individuals to apply to their daily lives for improved performance Stress Solutions provides individuals with opportunities to extend the SMART principles to domains of stress and resilience.
  Interventions: Behavioral: Strategic Memory Advanced Reasoning Training teaches meta-cognitive strategies for individuals to apply to their daily lives for improved performance

INTERVENTIONS:
Behavioral: Strategic Memory Advanced Reasoning Training teaches meta-cognitive strategies for individuals to apply to their daily lives for improved performance — Online SMART is a curriculum that teaches strategies of how to use the brain better, in such a way that may improve brain health and performance. SMART strives to achieve optimal cognitive function realized by the brain's ability to efficiently manage complex information by abstracting its essential meaning rather than attempting to memorize details, and to prioritize the information in order to attend to the most relevant parts.
  Stress Solutions extends the SMART principles to relevant domains of stress and resilience.
  Other Names: SMART

SUMMARY:
The combination of transcranial magnetic stimulation (TMS) and electroencephalography (EEG) has been suggested as a promising brain imaging tool for identifying biomarkers of brain health.

In this pilot study, study investigators will explore the neurophysiological metrics of brain health with a non-invasive brain imaging technique, alongside behavioral and fMRI metrics collected through another study (NCT04869111).

DETAILED DESCRIPTION:
The Direct Electro-Physiological Imaging medical device (Delphi-MD), developed by QuantalX Neuroscience, combines both TMS and EEG technologies. This is a non-invasive technique that uses magnetic pulses to temporarily stimulate specific brain areas in participants, and the EEG device records brain electrophysiological response to the stimulation.

Recruitment for this pilot study will be restricted to participants in the imaging cohort of a separate study, The BrainHealth Project (NCT04869111). As that cohort is already completing behavioral and fMRI metrics, this exploratory study would allow study investigators to examine relevant associations between those metrics with the neurophysiological metrics from the Delphi device.

Study participants will complete two in-person sessions with the Delphi-MD device that align with their pre-scheduled imaging appointments.

ELIGIBILITY:
Inclusion Criteria:

* Must be an active brain imaging participant in The BrainHealth Project (NCT04869111)
* Minimum age of 22
* Fluent in English
* Able to read & hear information over a computer
* Must pass an MRI safety screener to assess the presence of contraindicators for MRI compatibility (i.e., non-removable metal within/on the body, claustrophobia, pregnancy, non-correctable vision problems, head trauma, and CNS disease)or other standard requirements as determined by the Imaging Center.
* Must pass a modified TMS Adult Safety Screen
* Meet all criteria for study as determined by the study physician

Exclusion Criteria:

* A diagnosis of a neurodegenerative disease
* A history of stroke, concussion, or brain injury that currently hinders them from functioning at their prior level
* A diagnosis of autism spectrum disorder that currently hinders them from functioning independently.
* Metallic brain implants or fragments (like a shunt, pacemaker, clips, coils, bullet fragments, cochlear implants)
* Magnetically activated implants or electronically implanted devices
* Medication pumps
* Personal or family history of epilepsy, seizure(s), seizure disorder.
* History of, or risk factors for syncope (fainting)
* Report significant cognitive challenges
* Report untreated health issues (like substance abuse, hypertension, hypo- or hyper-thyroidism)
* Have claustrophobia

Ages: 22 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2025-09-03 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Correlation of DELPHI-MD Output Measures with the online BrainHealth Index | Up to one year
  Evaluate the strength and significance of correlations between DELPHI-MD output metrics (e.g., cortical excitability, local/global mean field potentials, response amplitude, and latency) and scores from the BrainHealth Index. Unit of Measurement: Correlation coefficient (r).
  (Minimum value: -1.0, Maximum value: 1.0) (Higher value represents stronger correlation)

SECONDARY OUTCOMES:
Correlation of DELPHI-MD Output Measures with Quantitative fMRI Metrics | Up to one year
  Assess the relationships between DELPHI-MD output metrics and the following fMRI metrics collected in separate study (i) functional connectivity, (ii) cerebral blood flow, (iii) cerebrovascular reactivity, and (iv) white matter integrity. Unit of Measurement: Correlation coefficient (r).
  (Minimum value: -1.0, Maximum value: 1.0) (Higher value represents stronger correlation)

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Chapman, PhD, Principal Investigator — The University of Texas at Dallas
Locations (1):
- Center for BrainHealth at The University of Texas at Dallas, Dallas, Texas, United States

REFERENCES:
- [Background] Rossi S, Antal A, Bestmann S, Bikson M, Brewer C, Brockmoller J, Carpenter LL, Cincotta M, Chen R, Daskalakis JD, Di Lazzaro V, Fox MD, George MS, Gilbert D, Kimiskidis VK, Koch G, Ilmoniemi RJ, Lefaucheur JP, Leocani L, Lisanby SH, Miniussi C, Padberg F, Pascual-Leone A, Paulus W, Peterchev AV, Quartarone A, Rotenberg A, Rothwell J, Rossini PM, Santarnecchi E, Shafi MM, Siebner HR, Ugawa Y, Wassermann EM, Zangen A, Ziemann U, Hallett M; basis of this article began with a Consensus Statement from the IFCN Workshop on "Present, Future of TMS: Safety, Ethical Guidelines", Siena, October 17-20, 2018, updating through April 2020. Safety and recommendations for TMS use in healthy subjects and patient populations, with updates on training, ethical and regulatory issues: Expert Guidelines. Clin Neurophysiol. 2021 Jan;132(1):269-306. doi: 10.1016/j.clinph.2020.10.003. Epub 2020 Oct 24. PMID 33243615
- [Background] Chapman SB, Fratantoni JM, Robertson IH, D'Esposito M, Ling GSF, Zientz J, Vernon S, Venza E, Cook LG, Tate A, Spence JS. A Novel BrainHealth Index Prototype Improved by Telehealth-Delivered Training During COVID-19. Front Public Health. 2021 Mar 16;9:641754. doi: 10.3389/fpubh.2021.641754. eCollection 2021. PMID 33796498
- [Background] Arrenberg AB, Driever W. Integrating anatomy and function for zebrafish circuit analysis. Front Neural Circuits. 2013 Apr 23;7:74. doi: 10.3389/fncir.2013.00074. eCollection 2013. PMID 23630469
- [Background] Zaghi S, Acar M, Hultgren B, Boggio PS, Fregni F. Noninvasive brain stimulation with low-intensity electrical currents: putative mechanisms of action for direct and alternating current stimulation. Neuroscientist. 2010 Jun;16(3):285-307. doi: 10.1177/1073858409336227. Epub 2009 Dec 29. PMID 20040569
- [Background] Rossini PM, Burke D, Chen R, Cohen LG, Daskalakis Z, Di Iorio R, Di Lazzaro V, Ferreri F, Fitzgerald PB, George MS, Hallett M, Lefaucheur JP, Langguth B, Matsumoto H, Miniussi C, Nitsche MA, Pascual-Leone A, Paulus W, Rossi S, Rothwell JC, Siebner HR, Ugawa Y, Walsh V, Ziemann U. Non-invasive electrical and magnetic stimulation of the brain, spinal cord, roots and peripheral nerves: Basic principles and procedures for routine clinical and research application. An updated report from an I.F.C.N. Committee. Clin Neurophysiol. 2015 Jun;126(6):1071-1107. doi: 10.1016/j.clinph.2015.02.001. Epub 2015 Feb 10. PMID 25797650
- [Background] Hallett M. Transcranial magnetic stimulation: a primer. Neuron. 2007 Jul 19;55(2):187-99. doi: 10.1016/j.neuron.2007.06.026. PMID 17640522
- [Background] Casarotto S, Romero Lauro LJ, Bellina V, Casali AG, Rosanova M, Pigorini A, Defendi S, Mariotti M, Massimini M. EEG responses to TMS are sensitive to changes in the perturbation parameters and repeatable over time. PLoS One. 2010 Apr 22;5(4):e10281. doi: 10.1371/journal.pone.0010281. PMID 20421968
- [Background] Lioumis P, Kicic D, Savolainen P, Makela JP, Kahkonen S. Reproducibility of TMS-Evoked EEG responses. Hum Brain Mapp. 2009 Apr;30(4):1387-96. doi: 10.1002/hbm.20608. PMID 18537115
- [Background] Fogel H, Levy-Lamdan O, Zifman N, Hiller T, Efrati S, Suzin G, Hack DC, Dolev I, Tanne D. Brain Network Integrity Changes in Subjective Cognitive Decline: A Possible Physiological Biomarker of Dementia. Front Neurol. 2021 Aug 30;12:699014. doi: 10.3389/fneur.2021.699014. eCollection 2021. PMID 34526957
- [Background] Levy-Lamdan O, Zifman N, Sasson E, Efrati S, Hack DC, Tanne D, Dolev I, Fogel H. Evaluation of White Matter Integrity Utilizing the DELPHI (TMS-EEG) System. Front Neurosci. 2020 Dec 21;14:589107. doi: 10.3389/fnins.2020.589107. eCollection 2020. PMID 33408607
- [Background] Maidan I, Zifman N, Hausdorff JM, Giladi N, Levy-Lamdan O, Mirelman A. A multimodal approach using TMS and EEG reveals neurophysiological changes in Parkinson's disease. Parkinsonism Relat Disord. 2021 Aug;89:28-33. doi: 10.1016/j.parkreldis.2021.06.018. Epub 2021 Jun 29. PMID 34216938
- [Background] Zifman N, Levy-Lamdan O, Suzin G, Efrati S, Tanne D, Fogel H, Dolev I. Introducing a Novel Approach for Evaluation and Monitoring of Brain Health Across Life Span Using Direct Non-invasive Brain Network Electrophysiology. Front Aging Neurosci. 2019 Sep 9;11:248. doi: 10.3389/fnagi.2019.00248. eCollection 2019. PMID 31551761